CLINICAL TRIAL: NCT04755673
Title: Open-Label Assessment of the Efficacy of Atrantil In the Treatment of Methane-Predominate Intestinal Bacterial Overgrowth
Brief Title: Atrantil for Intestinal Bacterial Overgrowth
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Northwestern University (Other)
Responsible Party: Principal Investigator, Darren Brenner, Associate Professor of Medicine and Surgery, Northwestern University
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Other
Other Study IDs: STU00212557
Record Dates: First submitted 2021-02-02; First posted 2021-02-16 (Actual); Last update posted 2023-01-12 (Actual); Status verified 2023-01

CONDITIONS: Irritable Bowel Syndrome; Bacterial Overgrowth Syndrome; SIBO
MeSH Terms: conditions — Irritable Bowel Syndrome; Blind Loop Syndrome

STUDY DESIGN:
Intervention Model Description: All participants receive 4 weeks (28 days)supply of Atrantil- 2 capsules 3 times per day .
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Experimental: Atrantil (Medical Food) (Experimental): All participants in the trial will take two capsules of Atrantil three times a day for 28 days.
  Interventions: Other: Atrantil (Medical Food)

INTERVENTIONS:
Other: Atrantil (Medical Food) — All participants will be given 28 days supply of Atrantil. The impact of the intervention will be measured by daily symptom surveys as well as a hydrogen methane breath test administered at the end of the 28 days of treatment to identify if methane levels have changed.

SUMMARY:
Intestinal Bacterial Overgrowth (IBO) is a common functional condition due to excessive amounts of bacteria in the gastrointestinal tract. These bacteria ferment ingested food resulting in the production of hydrogen, methane, and carbon dioxide which subsequently can induce GI symptoms including abdominal pain, bloating, distention, diarrhea and constipation. Typically this condition is treated with antibiotics but for a portion of patients symptoms often recur. Recent work suggests that increased methane production may emanate from overgrowth of a specific type of archaebacteria, causing the aforementioned symptoms. However, no current therapies exist to treat this phenomenon. The investigators propose to trial the supplement Atrantil on patients with IMO in order to study the supplements impact on symptoms, quality of life, and methane levels.

DETAILED DESCRIPTION:
Intestinal microbial overgrowth is associated with multiple gastrointestinal symptoms. Most prevalent are gas-related symptoms (i.e. bloating, distention, increased flatus, constipation)

. Intestinal microbial overgrowth can currently be divided into two main subcategories: small intestinal bacterial overgrowth (SIBO) and intestinal methanogenic overgrowth (IMO). Both are most commonly detected via breath testing-a simple non-invasive study

* Despite the increasing prevalence of this disorder few evidence-based therapeutics currently exist. SIBO, identified by elevations in breath hydrogen, has been shown to respond to treatment with antibiotics including rifaximin and doxycycline in clinical trials
* However, IMO, detected by elevations in breath methane is a different disorder attributed to overgrowth of archaea which reside predominately in the colon
* Currently, there are no evidence-based treatments for IMO, and the American College of Gastroenterology guideline on the diagnosis and treatment of SIBO makes no specific recommendations regarding the treatment of this disorder.

Atrantil is a medical food composed of peppermint, quebracho tree bark, and horse chestnut.

These components are purported to reduce methane production, scavenge hydrogen (thus reducing the building blocks for methane), and potentially act as a cidal agent for methanogenic archaea. In a small randomized controlled-trial, Atrantil reduced bloating and constipation in a population of individuals with irritable bowel syndrome with constipation (IBS-C)

Given these initial results the investigators hypothesize that Atrantil may represent an inexpensive and safe treatment for patients with excessive methane production. Thus, the purpose of this study is to determine whether the holistic treatment, Atrantil, is beneficial for the treatment of IMO.

ELIGIBILITY:
Inclusion Criteria:

1. Participants must be able to provide informed consent
2. Participants must be able to attend study visits
3. Participants aged 18 years or greater
4. Must have a diagnosis of Intestinal Methane Overgrowth based on North American Consensus/American College of Gastroenterology established cutoffs
5. Participants must report current symptoms of bloating, distention, abdominal pain, abdominal discomfort and constipation
6. Participant must be an established patient at Northwestern Memorial Hospital

Exclusion Criteria:

1. Participants who are already taking Atrantil
2. Participants who are pregnant or breast-feeding
3. Participants who cannot tolerate or are unwilling to complete a hydrogen-methane breath test at week 4.
4. Inability to attend all study visits and complete survey data.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 40 (Actual)
Dates: Start 2020-09-18 (Actual); Primary Completion 2022-09-26 (Actual); Study Completion 2022-09-27 (Actual)

PRIMARY OUTCOMES:
Change in clinical symptoms of Intestinal Methane Overgrowth as measured by daily Numeric Rating Scale (NRS) measuring pain, bloating, distention, and discomfort. | Daily for 28 days
  Numeric Rating Scale is a four-item scale measuring the severity of pain, bloating, distention, and discomfort on a scale of 1 to 10 for each measure. Higher scores indicate a higher level of symptom severity. Lower scores indicate a lower level of symptom severity.
Change in clinical symptoms of Intestinal Methane Overgrowth as measured by Patient Reported Outcome Measures Information Systems Gastrointestinal Symptoms Scale (PROMIS-GI) | Change from Baseline at four weeks.
  PROMIS GI Scales is a collection of eight categories of GI-symptoms (Belly pain, Bowel Incontinence, Constipation, Diarrhea, Disrupted Swallowing, Gas and Bloating, Nausea and Vomiting, and Acid reflux) Higher scores indicate a higher level of symptom severity. Lower scores indicate a lower level of symptom severity.
Change in clinical symptoms of Intestinal Methane Overgrowth as measured by the Bristol Stool Scale (BSS) | Change from Baseline at four weeks.
  BSS is a clinical tool that divides feces into 7 categories along the continuum severe constipation to severe diarrhea to demonstrate the effectiveness of a treatment

SECONDARY OUTCOMES:
Change in quality of life as measured by Short Form- 12. | Change from Baseline at four weeks.
  SF-12 scale is a generic, multipurpose short-form survey with 12 questions selected from the SF-36 Health Survey to evaluate overall health-related quality of life. Answers are combined, scored and weighted into mental and physical functioning component scales. The scores for each scale range from 0 to 100. A higher value indicates a better quality of life of the patient.
Change in Quality of life as measured by the PROMIS-Global Health (PROMIS-GH) | Change from Baseline at four weeks.
  PROMIS® Global Health Short Form (10 items). The 10 global health items include ratings of the five core PROMIS domains. It includes the most widely used self-rated health item (global01). PROMIS® includes a single item that provides a pure rating of physical health (global03) and another item for mental health (global04). Also included is an overall quality of life item (global02). The remaining items provide global ratings of physical function (global06), fatigue (global08), pain (global07), emotional distress (global10), and social health (global05 and global09). The 10 PROMIS® Global Health items each have 5 response choices, with the exception of the common 11-point pain intensity item ("How would you rate your pain on average" with 0=No pain and 10=Worst imaginable pain). Global 1-5, 9 range from 5 (Excellent) to 1 (Poor), with higher numbers meaning greater health. Certain items are restored (Global 7 such that 5=0 no pain, and 1=10 worst pain), Global8 (5=None, 1=Very Severe),
Change in methane as measured by hydrogen methane breath-test pre and post-treatment. | Post-Treatment (+-3 days)
  Methane levels equal to or more than 10 parts per million are considered abnormal and positive for intestinal methane overgrowth. Methane levels under 10 are considered normal and negative for intestinal methane overgrowth.

CONTACTS AND LOCATIONS:
Overall Officials: Darren Brenner, MD, Principal Investigator — Northwestern Memorial Hospital/Feinberg School of Medicine
Locations (1):
- Northwestern Medicine Digestive Health Center, Chicago, Illinois, United States

IPD SHARING:
Plan to Share IPD: No